CLINICAL TRIAL: NCT04494412
Title: An Open Label, Single Arm Study to Evaluate Single and Multiple Dose Pharmacokinetics, Safety and Tolerability, and to Explore Clinical Outcomes of Treatment With Intravenous (IV) Zanamivir in Neonates and Infants Under 6 Months of Age With Confirmed Complicated Influenza Infection
Brief Title: An Intravenous (IV) Zanamivir Pharmacokinetics (PK) Study in Hospitalized Neonates and Infants With Influenza Infection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200925
Record Dates: First submitted 2020-07-15; First posted 2020-07-31 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Influenza, Human; Arthralgia
Keywords: Human influenza; Zanamivir; Pediatric; Hospitalized neonates and infants
MeSH Terms: conditions — Influenza, Human; Arthralgia | interventions — Zanamivir

STUDY DESIGN:
Intervention Model Description: Open-label, multi-center and single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hospitalized neonates and infants with influenza infection (Experimental): Preterm neonates and infants who have reached Post-Menstrual Age (PMA) of at least 28 weeks and have a confirmed complicated influenza infection will be included. Participants will receive daily IV infusion of zanamivir for up to 5 days. This initial 5-day treatment course may be extended for up to 5 additional days if clinical symptoms, participant characteristics or virological tests warrant further treatment. The initial dose of IV zanamivir will be determined by PMA/corrected age and body weight. The maintenance dose and interval between the initial dose and subsequent twice-daily maintenance dose will be further determined by Principal Investigator based on renal function.
  Interventions: Drug: Zanamivir

INTERVENTIONS:
Drug: Zanamivir — Zanamivir solution for infusion will be available as a 10 milligrams per milliliters (mg/mL) vial. DECTOVA is approved for age groups 6 months and above.
  Other Names: DECTOVA

SUMMARY:
Influenza infection is an important public health priority, with seasonal outbreaks and pandemics causing considerable global morbidity and mortality. The PK, pharmacodynamics (PD), safety and efficacy of IV zanamivir have been evaluated in adults, adolescents and infants more than or equal to (>=) 6 months of age with hospitalized influenza in the IV zanamivir global development program. However, antiviral treatment of neonates and infants under 6 months of age hospitalized with influenza infection remains a medical unmet need. Given the immaturity of the immune system at this age, there are no licensed influenza vaccines for children aged less than six months old. As a requirement of the Pediatric Investigation Plan European Union (EU), GlaxoSmithKline (GSK) will be conducting this open-label, multi-center, single arm, post-marketing authorization study to evaluate the PK and collect safety and tolerability information of IV zanamivir in hospitalized neonates and infants under 6 months of age with confirmed complicated influenza infection. The total duration of study participation for each participant will be up to 24 days with a study treatment period up to 10 days and 14 days of post-treatment follow up. However, for a given participant, the initial 5-day treatment course may be extended for up to 5 additional days if clinical symptoms, participant characteristics or virological tests as assessed by the investigator warrant further treatment. DECTOVA is a trademark of GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants who are aged less than 6 months (corrected age) at the time of the informed consent signed by legally acceptable representative (LAR) of minors. Preterm neonates and infants will be eligible for inclusion but must have reached PMA of at least 28 weeks.
* Participants who are hospitalized with influenza infection, confirmed by a positive rapid molecular diagnostic test for influenza, or a local quantitative Reverse transcriptase-polymerase chain reaction (RT-PCR) test and who must have a potential for improvement Participants with negative rapid molecular test result suspected of having influenza can be enrolled following confirmatory testing by quantitative RT-PCR.
* Participants with a high risk of altered oral drug absorption, represented by multi-organ dysfunction (dysfunction of at least 2 organs, as defined by the treating physician). (applicable only for Netherlands)
* Body weight >=1 kilograms (kg).
* No gender restriction.
* LAR of minors are willing and able to give written informed consent to participate in the study (or included as permitted by local regulatory authorities, Independent Ethics Committees [IECs] or local laws).

Exclusion criteria:

* Participants who are known or suspected to be hypersensitive to any component of the study medication.
* Participants with a disease process which is likely to be irreversible.
* Liver function:

  * Participants who meet the following criteria at Baseline:

    1. Alanine transaminase (ALT) >=3 times upper limit of normal (ULN) with bilirubin >=2 times ULN
    2. or isolated bilirubin >=2 times ULN and >50 percent (%) direct bilirubin
    3. or ALT >=5 times ULN Inclusion of participants with liver function tests that fall outside these criteria must be discussed and agreed with the medical monitor.
  * Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of benign conditions such as Gilbert's syndrome). Inclusion of participants with neonatal hyperbilirubinemia may be considered if appropriately managed according to local guidelines and must be discussed with the medical monitor (Not-applicable for Great Britain).
* Participants who require concurrent therapy with another anti influenza drug.
* Participants who have participated in a study using an investigational drug within 30 days prior to Baseline.
* Child in care (CiC), as defined below:

  * A child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation.
  * The definition of a CiC can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a CiC does not include a child who is adopted or has an appointed legal guardian.
* Participants undergoing treatment by Extracorporeal membrane oxygenation (ECMO) or hemofiltration.
* Participants who are positive for severe acute respiratory syndrome-related coronavirus-2 (SARS-CoV-2) as determined by a diagnostic test, at screening

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve (AUC) of zanamivir | Up to 12 hours after end of infusion on Day 1
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of zanamivir.
Maximum observed serum concentration (Cmax) of zanamivir | Up to 12 hours after end of infusion on Day 1
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of zanamivir.
Clearance (CL) in plasma following administration of zanamivir | 30 minutes, 2 hours, 6 hours, 12 hours post dose on Day 1; predose on Days 3, 4 or 5
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of zanamivir.
Terminal half-life (t1/2) of zanamivir | 30 minutes, 2 hours, 6 hours, 12 hours post dose on Day 1; predose on Days 3, 4 or 5
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of zanamivir.

SECONDARY OUTCOMES:
Number of participants with adverse event(s) (AE) and serious adverse event(s) (SAE) | From start of treatment (Day 1) up to Day 24
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence resulting in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect or any other important medical event that may jeopardize the participant or may require medical or surgical treatment to prevent one of the other outcomes listed before.
Number of participants with abnormal findings in heart rate | From start of treatment (Day 1) up to Day 24
  Number of participants with abnormal findings for heart rate will be assessed.
Number of participants with abnormal findings in Oxygen Saturation | From start of treatment (Day 1) up to Day 24
  Number of participants with abnormal findings for Oxygen Saturation will be assessed.
Number of participants with abnormal findings in respiration rate | From start of treatment (Day 1) up to Day 24
  Number of participants with abnormal findings for respiration rate will be assessed.
Number of participants with abnormal findings in body temperature | From start of treatment (Day 1) up to Day 24
  Number of participants with abnormal findings for body temperature will be assessed.
Viral load over time after administration of zanamivir | Day 1 up to Maximum Day 24
  Nasopharyngeal swab samples will be collected for assessing quantitative viral load.
Change From Baseline in viral load after administration of zanamivir | Baseline (Day 1) and up to maximum Day 24
  Nasopharyngeal swab samples will be collected for assessing quantitative viral load.
Number of participants with phenotypic resistance | Up to Day 24
  Nasopharyngeal swab samples will be collected for assessing phenotypic resistance.
Number of participants with genotypic resistance | Up to Day 24
  Nasopharyngeal swab samples will be collected for assessing genotypic resistance.
Number of participants with emergence of resistance to zanamivir | Up to Day 24
  Nucleotide sequence analysis will be carried out to determine emergence of resistance to zanamivir.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Italy (4):
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Messina
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Roma
- GSK Investigational Site, Bydgoszcz, Poland
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/